CLINICAL TRIAL: NCT01735565
Title: Neutrophil Extracellular Trap Formation in Patients Undergoing Bone Marrow Transplant
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 56286
Record Dates: First submitted 2012-11-22; First posted 2012-11-28 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Bone Marrow Transplant
Keywords: NET formation; neutraphil extracellular traps; post-engraftment immune system

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post bone marrow transplant: Patients who are undergoing bone marrow transplant, as well as patients who have completed a bone marrow transplant within the previous year.

SUMMARY:
This is a prospective observational study to determine the point after bone marrow transplant in adults and children at which the neutrophils derived from the transplanted stem cells are competent to form functional neutrophil extracellular traps (NETs). Furthermore, given the importance of platelet function for NET formation, we also plan to examine platelet activation and function as well as the platelet transcriptome using the same clinical samples.

DETAILED DESCRIPTION:
Background and Introduction

The role of the human polymorphonuclear leukocytes (PMNs) in the acute inflammatory response is well documented. PMNs play a fundamental role in the innate immune response and are rapidly recruited to areas of injury or inflammation where they participate in bacterial phagocytosis and killing. Disorders associated with a deficiency or impairment of PMN function (neutropenia, chronic granulomatous disease (CGD), leukocyte adhesion deficiency) predispose to infections with bacteria and fungi. Regulation of this potent component of the acute inflammatory response is imperative to prevent overwhelming infections often associated with morbidity and mortality.

Recently, neutrophils isolated from healthy adult donors were shown to undergo programmed cell death distinct from apoptosis and necrosis to form neutrophil extracellular traps (NETs). NETs are extensive lattices of extracellular DNA and chromatin decorated with anti-microbial proteins and degradative enzymes such as myeloperoxidase and neutrophil elastase (NE). NETs effect extracellular killing of bacteria and fungi. The laboratory of Christian Yost, MD recently characterized impaired NET formation as a novel innate immune deficiency of human newborn infants and showed that PMNs isolated from the cord blood of newborn infants, both term and preterm, demonstrated impaired NET formation and extracellular bacterial killing as compared to PMNs isolated from healthy adults. However, the timing for developmental maturation of newborn infant PMN NET formation remains unknown.

Stem cells for bone marrow transplants originate from cord blood, peripheral stem cells, or bone marrow stem cells. Regardless of the source of these stem cells, patients receiving a bone marrow transplant are essentially building a new immune system, as if they were a newborn baby. Immune system reconstitution is a continuous process whose components can take up to 1 to 2 years to fully recover. Severe infections in bone marrow transplant patients occur and may be associated with deficient PMN NET formation by way of impaired extracellular bacterial containment and killing. We hypothesize that the increased risk of infection attributed to bone marrow transplant recipients results, in part, from deficient PMN NET formation by the nascent, post-engraftment immune system which is molecularly and functionally similar to that of a newborn baby. We plan to determine the point after transplant at which the neutrophils derived from the transplanted stem cells are competent to form functional NETs. Furthermore, given the importance of platelet function for NET formation, we also plan to examine platelet activation and function as well as the platelet transcriptome using the same clinical samples.

ELIGIBILITY:
Inclusion Criteria:

* Within one year of bone marrow transplant
* Informed consent

Exclusion Criteria:

* No specific exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are undergoing bone marrow transplant, as well as patients who have completed a bone marrow transplant within the previous year at Huntsman Cancer Institute and Primary Children's Medical Center will be identified as possible participants.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Post-engraftment maturation of NET formation | 1 year
  The time to post-engraftment maturation of NET formation capability in PMNs isolated from pediatric and adult patients undergoing bone marrow transplantation will be measured by serial blood sampling/analysis over the course of a year after transplant.

SECONDARY OUTCOMES:
Post-engraftment platelet function | 1 year
  Post-engraftment platelet function, transcriptome, and their potential influence on NET formation by PMNs will be measured by serial blood sampling/analysis over the course of a year after transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Yost, MD, Principal Investigator — University of Utah
Locations (3):
- United States (3):
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Primary Children's Medical Center, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Dinauer MC, Lekstrom-Himes JA, Dale DC. Inherited Neutrophil Disorders: Molecular Basis and New Therapies. Hematology Am Soc Hematol Educ Program. 2000:303-318. doi: 10.1182/asheducation-2000.1.303. PMID 11701548
- [Background] Brinkmann V, Reichard U, Goosmann C, Fauler B, Uhlemann Y, Weiss DS, Weinrauch Y, Zychlinsky A. Neutrophil extracellular traps kill bacteria. Science. 2004 Mar 5;303(5663):1532-5. doi: 10.1126/science.1092385. PMID 15001782
- [Background] Nathan C. Neutrophils and immunity: challenges and opportunities. Nat Rev Immunol. 2006 Mar;6(3):173-82. doi: 10.1038/nri1785. PMID 16498448
- [Background] Fuchs TA, Abed U, Goosmann C, Hurwitz R, Schulze I, Wahn V, Weinrauch Y, Brinkmann V, Zychlinsky A. Novel cell death program leads to neutrophil extracellular traps. J Cell Biol. 2007 Jan 15;176(2):231-41. doi: 10.1083/jcb.200606027. Epub 2007 Jan 8. PMID 17210947
- [Background] Buchanan JT, Simpson AJ, Aziz RK, Liu GY, Kristian SA, Kotb M, Feramisco J, Nizet V. DNase expression allows the pathogen group A Streptococcus to escape killing in neutrophil extracellular traps. Curr Biol. 2006 Feb 21;16(4):396-400. doi: 10.1016/j.cub.2005.12.039. PMID 16488874
- [Background] Urban CF, Reichard U, Brinkmann V, Zychlinsky A. Neutrophil extracellular traps capture and kill Candida albicans yeast and hyphal forms. Cell Microbiol. 2006 Apr;8(4):668-76. doi: 10.1111/j.1462-5822.2005.00659.x. PMID 16548892
- [Background] Bianchi M, Hakkim A, Brinkmann V, Siler U, Seger RA, Zychlinsky A, Reichenbach J. Restoration of NET formation by gene therapy in CGD controls aspergillosis. Blood. 2009 Sep 24;114(13):2619-22. doi: 10.1182/blood-2009-05-221606. Epub 2009 Jun 18. PMID 19541821
- [Background] Bianchi M, Niemiec MJ, Siler U, Urban CF, Reichenbach J. Restoration of anti-Aspergillus defense by neutrophil extracellular traps in human chronic granulomatous disease after gene therapy is calprotectin-dependent. J Allergy Clin Immunol. 2011 May;127(5):1243-52.e7. doi: 10.1016/j.jaci.2011.01.021. Epub 2011 Mar 3. PMID 21376380
- [Background] Yost CC, Cody MJ, Harris ES, Thornton NL, McInturff AM, Martinez ML, Chandler NB, Rodesch CK, Albertine KH, Petti CA, Weyrich AS, Zimmerman GA. Impaired neutrophil extracellular trap (NET) formation: a novel innate immune deficiency of human neonates. Blood. 2009 Jun 18;113(25):6419-27. doi: 10.1182/blood-2008-07-171629. Epub 2009 Feb 12. PMID 19221037
- [Background] Marcos V, Nussbaum C, Vitkov L, Hector A, Wiedenbauer EM, Roos D, Kuijpers T, Krautgartner WD, Genzel-Boroviczeny O, Sperandio M, Hartl D. Delayed but functional neutrophil extracellular trap formation in neonates. Blood. 2009 Nov 26;114(23):4908-11; author reply 4911-2. doi: 10.1182/blood-2009-09-242388. No abstract available. PMID 19965699
- [Background] Kraemer BF, Campbell RA, Schwertz H, Cody MJ, Franks Z, Tolley ND, Kahr WH, Lindemann S, Seizer P, Yost CC, Zimmerman GA, Weyrich AS. Novel anti-bacterial activities of beta-defensin 1 in human platelets: suppression of pathogen growth and signaling of neutrophil extracellular trap formation. PLoS Pathog. 2011 Nov;7(11):e1002355. doi: 10.1371/journal.ppat.1002355. Epub 2011 Nov 10. PMID 22102811
- [Background] Clark SR, Ma AC, Tavener SA, McDonald B, Goodarzi Z, Kelly MM, Patel KD, Chakrabarti S, McAvoy E, Sinclair GD, Keys EM, Allen-Vercoe E, Devinney R, Doig CJ, Green FH, Kubes P. Platelet TLR4 activates neutrophil extracellular traps to ensnare bacteria in septic blood. Nat Med. 2007 Apr;13(4):463-9. doi: 10.1038/nm1565. Epub 2007 Mar 25. PMID 17384648
- [Background] Rondina MT, Brewster B, Grissom CK, Zimmerman GA, Kastendieck DH, Harris ES, Weyrich AS. In vivo platelet activation in critically ill patients with primary 2009 influenza A(H1N1). Chest. 2012 Jun;141(6):1490-1495. doi: 10.1378/chest.11-2860. Epub 2012 Mar 1. PMID 22383669
- [Background] Rondina MT, Schwertz H, Harris ES, Kraemer BF, Campbell RA, Mackman N, Grissom CK, Weyrich AS, Zimmerman GA. The septic milieu triggers expression of spliced tissue factor mRNA in human platelets. J Thromb Haemost. 2011 Apr;9(4):748-58. doi: 10.1111/j.1538-7836.2011.04208.x. PMID 21255247
- [Background] Denis MM, Tolley ND, Bunting M, Schwertz H, Jiang H, Lindemann S, Yost CC, Rubner FJ, Albertine KH, Swoboda KJ, Fratto CM, Tolley E, Kraiss LW, McIntyre TM, Zimmerman GA, Weyrich AS. Escaping the nuclear confines: signal-dependent pre-mRNA splicing in anucleate platelets. Cell. 2005 Aug 12;122(3):379-91. doi: 10.1016/j.cell.2005.06.015. PMID 16096058